CLINICAL TRIAL: NCT01497704
Title: Evaluation of the Safety, Pharmacokinetics and Efficacy of Four Doses of YN968D1 in Subjects With Solid Tumors
Brief Title: Dose-Escalation and Safety Trial of YN968D1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Elevar Therapeutics (Industry)
Collaborators: Bukwang Pharmaceutical, Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BK-LSK-AM101; NCT01726101 (obsolete NCT alias)
Record Dates: First submitted 2011-12-18; First posted 2011-12-22 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Cancer Patients With Solid Tumors
Keywords: Cancer; Tumor; Oncology; Antiangiogenesis
MeSH Terms: conditions — Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- YN968D1 (Experimental): Active therapy arm for safety evaluation
  Interventions: Drug: YN968D1

INTERVENTIONS:
Drug: YN968D1 — Daily dosing of YN968D1 for treatment of solid tumors
  Other Names: Apatinib

SUMMARY:
This protocol will be divided into two parts: Part 1 will evaluate the safety and pharmacokinetics of three doses of YN968D1 after a single administration followed by a 28-Day continuous course of therapy; Part 2 will evaluate the safety and preliminary efficacy in an open-label administration of YN968D1 at the MTD or a maximum of 750 mg. All subjects in Part 1 and Part 2 of this study will be permitted to continue therapy with only safety monitoring and bimonthly assessments for progression, if the product is well tolerated and the subject has stable disease or better. Up to 72 subjects will be enrolled in this clinical trial.

DETAILED DESCRIPTION:
Part 1 will include a sequential evaluation of 3 subjects per cohort; cohort 1 at a dose of 100 mg YN968D1, followed by a cohorts 2, 3 and 4 at doses of 250 mg, 500 mg and 750 mg respectively. Initially, each subject will receive one dose of YN968D1 followed by a 7-Day observation period, during which single dose PK assessments and safety monitoring will be performed. If the initial dose is well tolerated, the subject will return on Day 8 and receive 28-Days of continuous YN968D1 oral administration daily. Each subject will subsequently be assessed for safety and disease progression on Day 35±2 and steady state pharmacokinetic sampling will be obtained. Patients may continue on therapy for an additional 28-Day cycles without dose interruption if the therapy is well tolerated. Efficacy assessments (biomarkers) and disease progression (RECIST imaging) will be assessed every two 28-Day cycles. The subjects will be assessed for safety for at least 28-Days after the last dose of YN968D1.

For Part 1 of this study, a Dose Limiting Toxicity (DLT) event is defined as any of the following events that are assessed by the Investigator as probably or possibly related to YN968D1 and occur during or after the initial dose on Day 1 through Day 35 of the first cycle of therapy.

* CTCAE Grade 4 event
* Grade 3 febrile neutropenia (<1,000 neutrophils/mL)
* Grade 3 hematologic toxicity with duration > 7 days
* Grade 3 non-hematologic toxicity (except for nausea, vomiting, diarrhea that continues despite optimal medical management)

If a DLT is experienced in any cohort, the cohort will be expanded to 6 subjects. If two (2) DLTs are experienced in any cohort, the study will be paused until the safety events are evaluated and discussed with the FDA to determine if the trial may continue.

Part 2 of this study will include up to 30 subjects. Each subject will receive a 750 mg dose or the maximum tolerated dose of YN968D1 from part 1 of the study for continuous 28-Day cycles of therapy. If a subject experiences an intolerable side effect a dose reduction or a dose interruption for up to 7-Days is allowed at the discretion of the investigator. Subjects will be evaluated for RECIST (version 1.1) response at the end of the second cycle of therapy on Day 56±3 of the Part 2 study. Safety reporting will be continued for 28-Days from the last dose of study medication.

All subjects in Part 1 and 2 of this trial will be eligible to continue therapy provided they have a least stable disease or better and are, in the opinion of the investigator, adequately tolerating treatment with YN968D1.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Subjects may be enrolled with the following malignancies:

   * Part 1: Subjects with any solid malignant tumor that are refractory to conventional therapy or the subject does not tolerate the conventional therapy
   * Part 2: Subjects diagnosed with NSCLC, CRC, RCC, Gastric cancer, GIST or triple negative Breast Cancer that are refractory to conventional therapy or the subject does not tolerate the conventional therapy
3. Evaluable disease defined by RECIST 1.1 as measured by a suitable imaging technique
4. Life expectancy ≥ 3 months
5. Subject must be suitable for oral administration of study medication
6. Signed written informed consent
7. Adequate bone marrow, renal, and liver function as manifested by the following:

   * CBC: ANC ≥ 1500/mm3, platelets ≥ 100,000/mm3, hemoglobin ≥ 9.0 g/dL
   * CMP: Creatinine clearance > 50 mL/min or serum creatinine < 1.5 x ULN, serum bilirubin < 2.5 x ULN, AST and ALT ≤ 5.0 × ULN
   * Coagulation profile with PT and INR, each ≤ 1.5 x ULN
   * Proteinuria < 200 mg by 24- hour urine collection without evidence of active sediment or hematuria
8. ECOG performance status ≤ 2
9. Female subjects of child-bearing potential must agree to use contraceptive measures starting 1 week before the administration of the first dose of YN968D1 until 4 weeks after discontinuing study drug and male subjects must agree to use contraceptive measures during the study and ending 4 weeks after last dose of study drug
10. Female patients of child-bearing potential are confirmed to have either a negative serum ß-hCG test, or have been evaluated by a gynecologist to confirm the patient is not pregnant, within 7 days prior to administration of initial dose of YN968D1
11. Ability and willingness to comply with the study protocol for the duration of the study and with follow-up procedures

Exclusion Criteria:

1. Pregnant or lactating women
2. Therapy with clinically significant systemic anticoagulant or antithrombotic agents within 7 days prior to first scheduled dose of YN968D1 that may prevent clotting and in the opinion of the investigator would place the subject at risk.
3. Hemoptysis within 3 months prior to first scheduled dose of YN968D1
4. Cytotoxic chemotherapy, immunotherapy, or radiotherapy within 4 weeks (6 weeks in cases of mitomycin C, nitrosourea, lomustine) prior to first scheduled dose of YN968D1
5. Surgery or visceral (e.g., hepatic or renal) biopsy within 28 days prior to first scheduled dose of YN968D1
6. Minor surgical procedure performed within 7 days prior to first scheduled dose of YN968D1
7. Prior exposure to YN968D1 (prior treatment with an angiogenesis inhibitor is not exclusionary)
8. Concomitant treatment with strong inhibitors or inducers of CYP3A4, CYP2C9 and CYP2C19.
9. Known history of human immunodeficiency virus infection (HIV)
10. Subjects with active bacterial infections and/or receiving systemic antibiotics
11. Current or past diagnosis of leukemia within the past 5 years
12. Prior radiotherapy at the target lesion
13. Known CNS metastases or clinical evidence of CNS involvement that is not stable for last 3 months by radiology documentation
14. Medical history of non-healing wound within past 2 weeks
15. History of bleeding diathesis or bleeding within 14 days prior to enrollment
16. Medical history of clinically significant thrombosis (bleeding or clotting disorder) within the past 3-months that in the opinion of the investigator may place the patient at risk of side effects on an anti-angiogenesis product
17. History of non-malignant GI bleeding, gastric stress ulcerations, or peptic ulcer disease within the past 3-months that in the opinion of the investigator may place the patient at risk of side effects on an anti-angiogenesis product
18. History of idiopathic or hereditary angioedema
19. History of sickle cell or any hemolytic anemia
20. History of uncontrolled hypertension that in the opinion of the investigator is not well managed by medication and may place the patient at risk when taking a VEGF inhibitor
21. Complete left bundle branch block (LBBB), bifascicular block (RBBB with either left anterior hemiblock or left posterior hemiblock)
22. Any clinically significant ST segment and/or T-wave abnormalities
23. Presence of unstable atrial fibrillation (ventricular response rate > 100 bpm). Patients with stable atrial fibrillation are allowed in the study provided they do not meet another exclusion criteria
24. Myocardial infarction or unstable angina pectoris within 6 months prior to starting study medication
25. Congestive heart failure (New York Heart Association class III-IV)
26. History of other significant cardiovascular disease or vesicular disease within the last 6 months (e.g. such as hypertensive crisis, hypertensive encephalopathy, stroke or TIA, or significant peripheral vascular disease) that in the opinion of the investigator may place the patient at risk when taking a VEGF inhibitor
27. History of significant gastrointestinal disorders that in the opinion of the investigator may place the patient at risk when taking a VEGF inhibitor; such as an abdominal fistula, GI perforation, or bleeding ulcer within 2 months of treatment
28. QTcF >450 msec on screening ECG
29. Baseline echocardiogram (within 2 months) with left ventricular ejection fraction (LVEF) <50%
30. History of clinically significant glomerulonephritis, biopsy proven tubulointerstitial nephritis, crystal nephropathy, or other renal insufficiencies
31. History of myocardial infarction within the past 6 months
32. Treatment with an investigational agent within the longest time frame of either 5 half-lives or 30 days of initiating study drug
33. Medical or psychiatric illness that, in the opinion of the Investigator, may impact the safety of the subject or objectives of the study
34. Known recreational substance use or psychiatric illness that, in the opinion of the Investigator, may affect compliance with scheduled visits
35. Known hypersensitivity to YN968D1 or components of the formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-04; Primary Completion 2015-02 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Safety in the first 28-Days of Therapy | 28-Days after Discontinuation of YN968D1
  The primary endpoint is evaluation of safety during the first 28-day cycle of therapy following the initiation of multiple dosing of YN968D1. The safety variables to be evaluated in this study are adverse events, physical examinations, vital signs (specifically including blood pressure), clinical laboratory evaluations including serum chemistry, hematology (including RBC morphology and reticulocyte count), and urinalysis (with detailed sediment analysis, proteinuria, and 24-hour urine for collection for creatinine clearance and protein), and electrocardiograms (ECGs) in triplicate.

SECONDARY OUTCOMES:
Pharmacokinetic Assessments for AUC, Cmax and Tmax | Day 1 Single Dose and Day 28 Steady State
  In Part 1 of this study, full PK profiles of YN968D1 will be obtained following administration of a single oral dose of YN968D1 on Day 1, and at steady state on Day 35±2. In Part 2 of this study, PK sampling will include a pre-dose and at the 4±1 hour time point on the first day of dosing in the first 28-Day cycle of therapy, and pre-dose on days 2, 7, 14 and 28 of the first 28-Day cycle of therapy
Tumor Biomarkers for Specific Tumor Types | Every 28-Days
  The primary Pharmacodynamic endpoints will include specific serum tumor markers for the target cancer, levels of endothelial growth factor (VEGF), and detection of EC-derived molecules such as sVEGFR-1, sVEGFR-2, sVEGFR-3, sTie-2 and VCAM-1, as well as PIGF. These biomarkers will be measured at baseline and at the end of every two 28-Day cycles of therapy. For patients that continue on repeat 28-Day cycles after the primary evaluation period, biomarkerts will be assessed after each two 28-Day cycles of therapy.
Objective Response Rate (RESIST) | Every 56-Days
  Anti-tumoral efficacy will be assessed by best radiographic response based on Response Evaluation Criteria in Solid Tumors (RECIST v 1.1) at baseline (Day -14 to -1) and at the end of two 28-Day cycles of therapy (Part 1 - Day 35±2; or Part 2 56±2 Days). For patients that continue on repeat 28-Day cycles after the primary evaluation period, progression will be assessed after each two 28-Day cycles of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Sharma, MD, FACP, Principal Investigator — Huntsman Cancer Institute; Yoon-Koo Kang, MD, PhD, Principal Investigator — Asan Medical Center
Locations (2):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States
- ASAN Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kang YK, Ryu MH, Hong YS, Choi CM, Kim TW, Ryoo BY, Kim JE, Weis JR, Kingsford R, Park CH, Jang S, McGinn A, Werner TL, Sharma S. Phase 1/2a Study of Rivoceranib, a Selective VEGFR-2 Angiogenesis Inhibitor, in Patients with Advanced Solid Tumors. Cancer Res Treat. 2024 Jul;56(3):743-750. doi: 10.4143/crt.2023.980. Epub 2024 Jan 18. PMID 38271925